CLINICAL TRIAL: NCT07317999
Title: Craniovertebral Angle and Neck Disability Among University Students With Forward Head Posture: A Comparative Study of Scapular Retraction Exercises Versus McKenzie Method
Brief Title: Effect of Scapular Retraction Exercises Versus McKenzie Method on CVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Forward Head Posture 0686
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Forward Head Posture; Craniovertebral Angle; Neck Disability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): scapular retraction exercises
  Interventions: Procedure: Scapular Retraction Exercises (SRE)
- 2 (Experimental): McKenzie method exercises
  Interventions: Procedure: McKenzie Method Exercises

INTERVENTIONS:
Procedure: Scapular Retraction Exercises (SRE) — Strengthen upper back muscles (scapular muscles, particularly the middle and lower trapezius and rhomboids) and improve posture.
  Arms: 1
Procedure: McKenzie Method Exercises — * Aim: Focus on self-treatment for neck pain and posture.
  * Duration: 20 minutes, 3 times a week
  Arms: 2

SUMMARY:
The goal of this quasi-experimental study is to compare the effectiveness of scapular retraction exercises versus the McKenzie method in improving craniovertebral angle (CVA), reducing neck pain, and minimizing neck disability among university students exhibiting forward head posture. The main question[s] it aims to answer [is/are]:

* Which of both exercises (scapular retraction or McKenzie method exercises) will be more effective in improvement craniovertebral alignment, alleviated pain, and decreased neck disability?

Group A performed scapular retraction exercises, while Group B practiced McKenzie method exercises. Both interventions were administered for 20 minutes, three times weekly over eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* University students with FHP
* Able to participate in exercise programs
* Free from severe musculoskeletal disorders or recent injuries

Exclusion Criteria:

* Students with contraindication to exercise,
* Individuals with neurological conditions affecting posture

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) | 8 weeks
  The angle is formed at the intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No